CLINICAL TRIAL: NCT04733976
Title: Assessing the Frequency and Experience of Bullying or Peer Victimization in Children With Muscular Dystrophy and Congenital Myopathies
Brief Title: Bullying in Youth With Muscular Dystrophy and Congenital Myopathies
Status: Completed | Type: Observational
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Laura McAdam, Physician, Holland Bloorview Kids Rehabilitation Hospital
Other Study IDs: McAdam_Bullying
Record Dates: First submitted 2021-01-22; First posted 2021-02-02 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Muscular Dystrophies; Congenital Myopathy
Keywords: muscular dystophy; congenital myopathy; youth; bullying; cyberbullying
MeSH Terms: conditions — Muscular Dystrophies; Myotonia Congenita; Bullying; Cyberbullying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bullying is an epidemic in Canada, and rates may be underreported. Youth with a disability were more likely to be bullied that those without disabilities, specifically if the disability was visible. Research has been conducted on the prevalence and effects of bullying in youth with disabilities such as cerebral palsy, obesity, and chronic pain; however, there is a paucity of research involving youth with muscular dystrophy and congenital myopathies. The objectives of this study are to: (1) measure bullying frequency, (2) describe the types of bullying experiences; and (3) explore barriers and facilitators to dealing with bullying by youth with muscular dystrophy or congenital myopathies and their parents. The objectives will be met by an online survey and qualitative interviews of youth with muscular dystrophy and congenital myopathy and their parents.

DETAILED DESCRIPTION:
Bullying is an epidemic in Canada. At least one in three Canadian youth report having been bullied. Bullying is defined as intentional aggressive behaviour with the intention to harm the victim. It is characterized by an imbalance of power between the perpetrator and the victim, and is often repetitive although it does not need to be. Studies have shown that youth with chronic illness or disability were more likely to be bullied that those without disabilities, specifically if the disability was visible. Research has been conducted on the prevalence and effects of bullying in youth with disabilities such as cerebral palsy, obesity, and chronic pain; however, there is a paucity of research involving youth with muscular dystrophy and congenital myopathies. The objectives of this study are to: (1) measure bullying frequency, (2) describe the types of bullying experiences; and (3) explore barriers and facilitators to dealing with bullying by youth and their parents. The objectives will be met using a cross-sectional, multi-centre, mixed methods approach. A survey will be administered online at a single time-point to youth and their parents. Then, purposefully selected participants and their parents will complete a qualitative interview.

ELIGIBILITY:
Inclusion Criteria:

* Muscular dystrophy or congenital myopathy diagnosis
* 10-19 years old
* Speaks and reads English or French

Exclusion Criteria:

* N/A

Ages: 10 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: Youth with a muscular dystrophy or congenital myopathy diagnosis from the neuromuscular clinics at the study sites (Holland Bloorview and CHEO) will be invited to participate in the study. The youth's parents will also be invited to participate with their child.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Demographics Form | Through study completion, 1 year
  This form was purposefully developed by the research team to capture characteristics such as age, gender, family demographics, schooling and academic success, muscular dystrophy or congenital myopathy diagnosis, comorbidities, physical function and mobility levels, and technology use. There is a participant version and a parent/guardian version.
Bullying and Cyberbullying: Perpetrators, Victims and Witnesses Survey (B&C:PVWS) | Through study completion, 1 year
  An amended version of the B&C:PVWS, developed by Mishna et al., to identify bullying and cyberbullying experiences of victims and perpetrators. The survey examines types of bullying experiences (e.g., physical, verbal, social, sexual), the context in which bullying occurs (e.g., race, sexual orientation, disability), and the participant's response to bullying and cyberbullying (e.g., sadness, actions taken, etc.). Perspectives on bullying and cyberbullying, as well as thoughts on potential interventions are sought. Questions measuring experiences of bully victimization and perpetration had good internal consistency with Cronbach alphas of .77 and .71, respectively.
Bullying Perspectives | Through study completion, 1 year
  A single question from The Bully Survey by Swearer et al. will be used to capture the youth participant's perspectives on bullying. They will be asked, "How much do you agree with each sentence?" on a 5-point scale (Totally false, somewhat false, both true and false, somewhat true, totally true).
PedsQL(TM) 3.0 Neuromuscular Module | Through study completion, 1 year
  The PedsQL(TM) 3.0 Neuromuscular Module assesses quality of life on three scales: 1) About my neuromuscular disease (17 items), 2) Communication (3 items), and 3) About our family resources (5 items). Participants are asked to indicate how much of a problem each of the statements has been for them on a 5-point Likert scale (0 = Never through 5 = Almost Always). Raw item scores are scaled linearly for a total score out of 100. As well, scale scores can be computed as an average of the total scale score. A higher score indicates better health-related quality of life (HRQoL). Two versions will be used in this study: Child Report (8-12 years old) and Teenager Report (13-18 years old), along with parent reports for each of these versions. All versions being used can be found in Appendix R. The child self-report has exemplary reliability (α = .85).
KIDSCREEN-10 Index | Through study completion, 1 year
  The KIDSCREEN-10 Index is a 10-item questionnaire developed to assess the HRQoL of children and young people 8-18 years old. Items in the questionnaire ask participants their thoughts on their health over the past week on a 5-point scale (Excellent, very good, good, fair, poor). Rasch analysis of raw scores provides a global unidimensional latent HRQoL score. Higher scores indicate better HRQoL. The KIDSCREEN-10 Index is reported to have good internal consistency (α = .82), and good test-retest reliability and stability (r = .73, ICC = .72).
EPOCH Measure of Adolescent Well-being (EPOCH) | Through study completion, 1 year
  The EPOCH assesses five positive psychological characteristics (i.e., engagement, perseverance, optimism, connectedness and happiness) that may facilitate the well-being, physical health and other positive outcomes in adulthood. Participants are instructed to indicate how much a statement describes them on a 5-point scale (Almost never, sometimes, often, very often, almost always). There are four items for each of the five domains. The EPOCH has exemplary overall reliability (α = .92).
Qualitative Interview | Through study completion, 1 year
  Participants will be purposefully selected to complete a semi-structured qualitative interview based on their survey results. Criteria for qualitative interview selection will be based on diversity of gender, school level, muscular dystrophy or congenital myopathy diagnosis, mobility, bullying and cyberbullying victimization, etc. Participants will be asked to describe specific bullying experiences, motivations, perspectives, and getting help.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molcho M, Craig W, Due P, Pickett W, Harel-Fisch Y, Overpeck M; HBSC Bullying Writing Group. Cross-national time trends in bullying behaviour 1994-2006: findings from Europe and North America. Int J Public Health. 2009 Sep;54 Suppl 2:225-34. doi: 10.1007/s00038-009-5414-8. PMID 19618108
- [Background] Pinquart M. Systematic Review: Bullying Involvement of Children With and Without Chronic Physical Illness and/or Physical/Sensory Disability-a Meta-Analytic Comparison With Healthy/Nondisabled Peers. J Pediatr Psychol. 2017 Apr 1;42(3):245-259. doi: 10.1093/jpepsy/jsw081. PMID 27784727
- [Background] Whitney DG, Peterson MD, Warschausky SA. Mental health disorders, participation, and bullying in children with cerebral palsy. Dev Med Child Neurol. 2019 Aug;61(8):937-942. doi: 10.1111/dmcn.14175. Epub 2019 Feb 1. PMID 30710352
- [Background] van Geel M, Vedder P, Tanilon J. Are overweight and obese youths more often bullied by their peers? A meta-analysis on the correlation between weight status and bullying. Int J Obes (Lond). 2014 Oct;38(10):1263-7. doi: 10.1038/ijo.2014.117. Epub 2014 Jul 8. PMID 25002148
- [Background] Fales JL, Rice S, Aaron RV, Palermo TM. Traditional and cyber-victimization among adolescents with and without chronic pain. Health Psychol. 2018 Mar;37(3):291-300. doi: 10.1037/hea0000569. Epub 2017 Nov 20. PMID 29154604
- [Background] Mishna F, McInroy LB, Lacombe-Duncan A, Bhole P, Van Wert M, Schwan K, Birze A, Daciuk J, Beran T, Craig W, Pepler DJ, Wiener J, Khoury-Kassabri M, Johnston D. Prevalence, Motivations, and Social, Mental Health and Health Consequences of Cyberbullying Among School-Aged Children and Youth: Protocol of a Longitudinal and Multi-Perspective Mixed Method Study. JMIR Res Protoc. 2016 May 24;5(2):e83. doi: 10.2196/resprot.5292. PMID 27220556
- [Background] Swearer SM, Cary PT. Perceptions and Attitudes Toward Bullying in Middle School Youth: A Developmental Examination Across the Bully/Victim Continuum. Journal of Applied School Psychology. 2003 Dec 12;19(2):63-79.
- [Background] Ravens-Sieberer U, Herdman M, Devine J, Otto C, Bullinger M, Rose M, Klasen F. The European KIDSCREEN approach to measure quality of life and well-being in children: development, current application, and future advances. Qual Life Res. 2014 Apr;23(3):791-803. doi: 10.1007/s11136-013-0428-3. Epub 2013 May 18. PMID 23686556
- [Background] Kern ML, Benson L, Steinberg EA, Steinberg L. The EPOCH Measure of Adolescent Well-Being. Psychol Assess. 2016 May;28(5):586-97. doi: 10.1037/pas0000201. Epub 2015 Aug 24. PMID 26302102
- [Background] Iannaccone ST, Hynan LS, Morton A, Buchanan R, Limbers CA, Varni JW; AmSMART Group. The PedsQL in pediatric patients with Spinal Muscular Atrophy: feasibility, reliability, and validity of the Pediatric Quality of Life Inventory Generic Core Scales and Neuromuscular Module. Neuromuscul Disord. 2009 Dec;19(12):805-12. doi: 10.1016/j.nmd.2009.09.009. Epub 2009 Oct 28. PMID 19846309
- See also: Common D, Singh A, Taylor C. "I thought he was dead": CBC survey reveals 4 in 10 boys are physically assaulted at school. CBC News. 2019 Oct 24. — http://www.cbc.ca/news/canada/school-violence-marketplace-1.5224865